CLINICAL TRIAL: NCT00545155
Title: Screening and Interventions in an Acute Care Setting
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Manish Shah, Professor, University of Rochester
Other Study IDs: AG028942-01; K23AG028942-01 (NIH)
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Results first posted 2012-09-28 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-05

CONDITIONS: Depression; Medication Administered in Error; Cognitive Impairment
MeSH Terms: conditions — Depression; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Geriatric EMS Patients: Cohort for reliability and concurrent validity testing.

SUMMARY:
The purpose of this study is to: 1) evaluate the reliability and validity of EMS screening for depression and cognitive impairment and 2) to develop a pilot ED intervention program to address the needs of older adults found to be at risk for depression and cognitive impairment.

DETAILED DESCRIPTION:
Many older adults (age over 64) have undetected health problems and lack basic prevention measures. Failure to identify and treat these conditions can lead to unnecessary morbidity and mortality and a decreased quality of life. Traditional screening and intervention programs, usually based in primary care providers' offices, have been insufficient, particularly in medically underserved populations. Alternate sites for screening and intervention have begun to receive attention and may hold promise.

The emergency medical services (EMS) system is a unique, community-wide system that can be used to perform in-home evaluations to uniformly screen large numbers of vulnerable older adults during emergency responses. The emergency department (ED) is the entry point for access to medical and social services for many patients. Recent programs have used the EMS system to screen patients or the ED to screen and intervene with mixed results, but little has been done to rigorously evaluate an integrated program of EMS screening that leads to focused ED interventions that promote the health of older adults. This proposed project builds upon the principal investigator's preliminary work and unique resources in Rochester, NY to develop and evaluate a program of EMS screening and ED interventions to help community-dwelling older adults with unmet needs. Specifically, this study aims to:

1. Implement an EMS screening program to identify community-dwelling older adults' unmet needs during emergency responses, identifying patients with needs related to depression and dementia.
2. Evaluate the test-retest reliability and concurrent criterion validity of EMS screening for depression and cognitive impairment.
3. Develop and refine an EMS and ED intervention program that addresses the needs of older adults found by EMS to be at risk for depression and cognitive impairment.

Upon completion, this study will have demonstrated the reliability and validity of EMS screening for these conditions and will have proposed an EMS and ED based intervention program template that can be applied to these and a wider range of geriatric disorders.

ELIGIBILITY:
Inclusion Criteria:

* age 65 or older, cared for by participating EMS providers

Exclusion Criteria:

* too ill to participate, not transported to participating hospitals

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Geriatric EMS patients
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2007-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manish N Shah, MD MPH, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Geriatric EMS Patients
Started | 187
Completed | 187
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Geriatric EMS Patients
Number analyzed (Participants) | 187
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.6 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120
  Male | 67
Region of Enrollment [Number; unit: participants]
  United States | 187

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Cognitively Impaired in Emergency Medical Services (EMS)
Description: Through testing using the Six Item Screener, this measure indicates the proportion of individuals cognitively impaired when tested by EMS personnel.
Time Frame: Upon testing by EMS.
Population: All of the subjects enrolled who completed follow up and completed all aspects of the testing.
Measure: Number; unit: percentage of subjects
Arm/Group | Geriatric EMS Patients
Number analyzed (Participants) | 186
percentage of subjects | 17 [4 to 25]

2. Primary Outcome: Proportion of Subjects Cognitively Impaired in the Emergency Department (ED)
Description: Through testing using the Six Item Screener, this measure indicates the proportion of individuals cognitively impaired when tested by study personnel in the ED.
Time Frame: Within 2 hours of testing by EMS.
Population: All of the subjects enrolled who completed all aspects of the testing.
Measure: Number; unit: percentage of subjects
Arm/Group | Geriatric EMS Patients
Number analyzed (Participants) | 186
percentage of subjects | 16

3. Primary Outcome: Proportion of Subjects Cognitively Impaired in the ED
Description: Through testing using the Mini-Cog, this measure indicates the proportion of individuals cognitively impaired when tested by study personnel.
Time Frame: Within 2 hours of testing by EMS
Population: All of the subjects enrolled who completed follow up and completed all aspects of the testing.
Measure: Number; unit: percentage of subjects
Arm/Group | Geriatric EMS Patients
Number analyzed (Participants) | 161
percentage of subjects | 55

4. Primary Outcome: Test-Retest Reliability of Six Item Screener Screening
Description: The Six Item Screener test for cognitive impairment (answer=yes or no)as performed by EMS personnel and study personnel.
Time Frame: 2 hours
Population: All of the subjects enrolled who completed follow up and completed all aspects of the testing.
Measure: Number (95% Confidence Interval); unit: kappa
Arm/Group | Geriatric EMS Patients
Number analyzed (Participants) | 186
kappa | 0.52 [0.36 to 0.69]

5. Primary Outcome: Concurrent Criterion Validity of Six Item Screener Screening
Description: This is the Six Item Screener test for cognitive impairment (scoring=yes or no), as compared to performing the Mini-Cog for cognitive impairment (scoring=yes or no) on patients immediately afterwards.
  This is concurrent criterion testing (two different instruments, neither being a gold standard) rather than the previous test-retest reliability testing (testing the same instrument twice).
Time Frame: 2 hours
Measure: Number (95% Confidence Interval); unit: kappa
Arm/Group | Geriatric EMS Patients
Number analyzed (Participants) | 187
kappa | 0.23 [0.13 to 0.34]

6. Primary Outcome: Proportion of Subjects Depressed in EMS.
Description: Through testing using the Patient Health Questionnaire-2 (PHQ-2), this measure indicates the proportion of individuals depressed when tested by EMS personnel
Time Frame: Upon testing by EMS.
Population: All of the subjects enrolled who completed follow up and completed all aspects of the testing.
Measure: Number; unit: percentage of subjects
Arm/Group | Geriatric EMS Patients
Number analyzed (Participants) | 178
percentage of subjects | 48 [19 to 38]

7. Primary Outcome: Proportion of Subjects Depressed in the ED
Description: Through testing using the PHQ-2, this measure indicates the proportion of individuals depressed when tested by study staff in the ED.
Time Frame: Within 2 hours of EMS testing.
Population: All of the subjects enrolled who completed follow up and completed all aspects of the testing.
Measure: Number; unit: percentage of subjects
Arm/Group | Geriatric EMS Patients
Number analyzed (Participants) | 179
percentage of subjects | 40

8. Primary Outcome: Proportion of Subjects Depressed in the ED
Description: Through testing using the PHQ-9, this measure indicates the proportion of individuals depressed when tested by study staff in the ED.
Time Frame: Within 2 hours of EMS testing
Population: All of the subjects enrolled who completed follow up and completed all aspects of the testing.
Measure: Number; unit: percentage of subjects
Arm/Group | Geriatric EMS Patients
Number analyzed (Participants) | 180
percentage of subjects | 22

9. Primary Outcome: Test-Retest Reliability Testing of PHQ-2 Screening
Description: The test for depression, using the PHQ-2, with scoring yes or no.
Time Frame: 2 hours
Measure: Number (95% Confidence Interval); unit: kappa
Arm/Group | Geriatric EMS Patients
Number analyzed (Participants) | 187
kappa | 0.50 [0.37 to 0.63]

10. Primary Outcome: Concurrent Criterion Validity of PHQ-2
Description: This is the PHQ-2, a test for depression (scoring=yes or no) as compared to the PHQ-9, a test for depression (scoring=yes or no), looking at the presence of depression.
  This is concurrent criterion testing (two different instruments, neither being a gold standard) rather than the previous test-retest reliability testing (testing the same instrument twice).
Time Frame: 2 hours
Measure: Number (95% Confidence Interval); unit: kappa
Arm/Group | Geriatric EMS Patients
Number analyzed (Participants) | 187
kappa | 0.36 [0.24 to 0.48]

ADVERSE EVENTS:
Arm/Group | Geriatric EMS Patients
Serious Adverse Events (participants affected / at risk) | 0/187
Other Adverse Events (participants affected / at risk) | 0/187

LIMITATIONS AND CAVEATS:
* administration of one measure was done by individuals not blinded to another, potentially improving the concurrent criterion validity results.
* a number of subjects did not consent or could not consent to participate in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No